CLINICAL TRIAL: NCT06748664
Title: A Clinical Trial of Rimegepant for Vestibular Migraine Evaluation: Pre-experiment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2024-0366
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-02

CONDITIONS: Vestibular Migraine; Adults 18 Years and Older (no Other Exclusion Criteria)
MeSH Terms: interventions — rimegepant sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A1:Rimegepant ODT 75mg, QD (Experimental)
  Interventions: Drug: Rimegepant
- Group A2: Placebo, QD (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rimegepant — Take 75mg qd of oral sulfate remigipan orally disintegrating tablets
  Arms: Group A1:Rimegepant ODT 75mg, QD
Drug: Placebo — Take 75mg qd of oral Rimegepan oral tablets with placebo
  Arms: Group A2: Placebo, QD

SUMMARY:
Vestibular migraine (VM) is one of the most common vestibular disorders, affecting 1.0% to 2.7% of the general population1, 7% of patients with definite migranous vertigo in dizziness clinics2, as well as 10.3% of VM patients in headache clinics3; 65% to 85% of VM patients are female1. Despite the relative prevalence of vestibular migraine, evidence-based medicine remains scarce. Two Cochrane reviews published in 2023 found that there is almost no evidence to support the use of medications for the acute treatment or preventive treatment of VM4,5.

Calcitonin gene-related peptide (CGRP) has been established as an excellent target for the treatment of migraine. Animal studies suggest a link between CGRP and vestibular disorders. A prospective observational cohort study found that monoclonal antibodies targeting CGRP receptors and ligands were very effective for vestibular migraine (VM), with 90% of participants experiencing at least a 50% reduction in vertigo attacks6. A small-scale prospective randomized controlled trial showed that a monoclonal antibody targeting a CGRP ligand significantly reduced the number of dizziness days per month in VM patients compared to placebo7. The efficacy of CGRP small molecule antagonists for the preventive and acute treatment of migraines has been widely recognized8,9. Therefore, we speculate that Rimegepant is effective for the preventive and acute treatment of vestibular migraine.

By focusing on a large sample RCT, our study can offer new evidence-based treatment options for patients with vestibular migraine. This is crucial, as many patients with vestibular migraine may not respond well to conventional migraine treatments. Our findings could guide clinicians in choosing more effective therapeutic strategies.

Specifically in acute treatment of vestibular migraine, triptans have failed to show superiority when compared to placebo in treatment vestibular migraine symptoms10. Prochlorperazine, a vestibular sedative, is widely used for acute treatment of vestibular migraine but is known to chronify symptoms11. Should rimegepant demonstrate superiority to placebo in this study, rimegepant could potentially become the first-line treatment for vestibular migraine across the world.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 years
* Documentation of a VM diagnosis according to the Barany Society/ ICHD-31
* More than 4 definite dizzy days per month in the 3 months prior to screen

  ≥1 prior preventive treatment failure
* E-diary compliance ≥ 80% during observational phase

Exclusion Criteria:

* Pregnant women, lactating women, or reluctance to use approved contraception during study participation;
* There is a condition or abnormality that the investigator believes will affect the safety of the patients or the quality of the data;
* Allergic to the ingredients of Remeipine sulfate or sulfate;
* Previous treatment with remejepam;
* History of ear surgery (except for ear tube surgery);
* Other vestibular diagnoses (excluding treated benign paroxysmal positional vertigo BPPV). Including Meniere's disease, superior semicircular canal prolapse syndrome, vestibular neuritis, persistent postural perceptual vertigo, unilateral or bilateral loss of vestibular function, cerebellar or brainstem disease, multiple sclerosis or sea sickness;
* Failure of more than 2 preventive migraine drugs;
* Previous or current treatment with CGRP drugs;
* History of serious medical or mental illness (including significant coronary artery disease, peripheral vascular disease, cerebrovascular disease, kidney disease, liver disease, Raynaud's disease, uncontrollable mental illness, or past psychiatric hospitalization, at the discretion of the treating physician);
* A history of mania, psychosis, or suicidal ideation;
* Acceptable if no more than two drugs for migraine prevention (prescribed specifically for this purpose) are used and the dose has stabilized for 2 months before the start of the study;
* History of drug or alcohol abuse based on the subject's medical record or self-reported report within 12 months before the screening period;
* Bototoxin (e. g., Dysport®, ®, Xeomin®, Myobloc®, and JeuveauTM) for the head, face, or neck during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | from baseline to weeks 12-16
  Change in number of Moderate/Severe vestibular symptom days as defined by Barany Society1 for participants measured daily from the observational phase compared to weeks 12-16.

SECONDARY OUTCOMES:
Secondary objectives for Preventive Treatment Group | every 4 weeks during the 12-week treatment period compared to baseline
  Change in number of Moderate/Severe vestibular symptom days as defined by Barany Society1 every 4 weeks during the 12-week treatment period compared to baseline
Secondary objectives for Preventive Treatment Group | every 4 weeks compared to baseline over the 12-week treatment period
  Change in the number of vestibular symptom attacks every 4 weeks compared to baseline over the 12-week treatment period. (Since VM attacks may recur multiple times within a day, each lasting a short duration, we need to further clearly define what constitutes "one attack.")
Secondary objectives for Preventive Treatment Group | every 4 weeks compared to baseline over the 12-week treatment period
  Change in the number of monthly migraine days (MMD) every 4 weeks compared to baseline over the 12-week treatment period
Secondary objectives for Preventive Treatment Group | from baseline to week 16
  Change in Migraine Disability Assessment (MIDAS) score from baseline to week 16
Secondary objectives for Preventive Treatment Group | from baseline to weeks 12-16
  Change in response rate (100%,75%,50%,25%,0%) by percentage reduction in moderate/severe vestibular symptom days from baseline to weeks 12-16
Secondary objectives for Preventive Treatment Group | from baseline to week 16
  Change in dizziness handicap inventory (DHI) score from baseline to week 16
Secondary objectives for Preventive Treatment Group | from baseline to week 16
  Change in Vestibular Activities of Daily Living Scale (VADL) score from baseline to week 16
Secondary objectives for Preventive Treatment Group | from baseline to week 16
  Change in Patient Health Questionnaire-9 (PHQ-9) score from baseline to week 16
Secondary objectives for Preventive Treatment Group | from baseline to week 16
  Change in General Anxiety Disorder-7 (GAD-7) score from baseline to week 16
Secondary objectives for Preventive Treatment Group | from baseline to week 16
  Change in Patient Global Impression of Change（PGIC scale）from baseline to week 16
Secondary objectives for Preventive Treatment Group | from baseline to week 16
  Change in Migraine-Specific Quality of Life (MSQ) score from baseline to week 16

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Croop R, Goadsby PJ, Stock DA, Conway CM, Forshaw M, Stock EG, Coric V, Lipton RB. Efficacy, safety, and tolerability of rimegepant orally disintegrating tablet for the acute treatment of migraine: a randomised, phase 3, double-blind, placebo-controlled trial. Lancet. 2019 Aug 31;394(10200):737-745. doi: 10.1016/S0140-6736(19)31606-X. Epub 2019 Jul 13. PMID 31311674
- [Background] Yu S, Kim BK, Guo A, Kim MH, Zhang M, Wang Z, Liu J, Moon HS, Tan G, Yang Q, McGrath D, Hanna M, Stock DA, Gao Y, Croop R, Lu Z. Safety and efficacy of rimegepant orally disintegrating tablet for the acute treatment of migraine in China and South Korea: a phase 3, double-blind, randomised, placebo-controlled trial. Lancet Neurol. 2023 Jun;22(6):476-484. doi: 10.1016/S1474-4422(23)00126-6. PMID 37210098
- [Background] Sharon JD, Krauter R, Chae R, Gardi A, Hum M, Allen I, Levin M. A placebo controlled, randomized clinical trial of galcanezumab for vestibular migraine: The INVESTMENT study. Headache. 2024 Nov-Dec;64(10):1264-1272. doi: 10.1111/head.14835. Epub 2024 Sep 30. PMID 39344988
- [Background] Russo CV, Sacca F, Braca S, Sansone M, Miele A, Stornaiuolo A, De Simone R. Anti-calcitonin gene-related peptide monoclonal antibodies for the treatment of vestibular migraine: A prospective observational cohort study. Cephalalgia. 2023 Apr;43(4):3331024231161809. doi: 10.1177/03331024231161809. PMID 36946234
- [Background] Webster KE, Dor A, Galbraith K, Haj Kassem L, Harrington-Benton NA, Judd O, Kaski D, Maarsingh OR, MacKeith S, Ray J, Van Vugt VA, Burton MJ. Pharmacological interventions for acute attacks of vestibular migraine. Cochrane Database Syst Rev. 2023 Apr 12;4(4):CD015322. doi: 10.1002/14651858.CD015322.pub2. PMID 37042545
- [Background] Webster K, Dor A, Galbraith K, Kassem LH, Harrington-Benton N, Judd O, Kaski D, Maarsingh O, MacKeith S, Ray J, Van Vugt V, Burton M. Pharmacological interventions for prophylaxis of vestibular migraine. Cochrane Database Syst Rev. 2023 Apr 12;2023(4):CD015187. doi: 10.1002/14651858.CD015187.pub2. PMID 37073858
- [Background] Cho SJ, Kim BK, Kim BS, Kim JM, Kim SK, Moon HS, Song TJ, Cha MJ, Park KY, Sohn JH. Vestibular migraine in multicenter neurology clinics according to the appendix criteria in the third beta edition of the International Classification of Headache Disorders. Cephalalgia. 2016 Apr;36(5):454-62. doi: 10.1177/0333102415597890. Epub 2015 Jul 29. PMID 26224714
- [Background] Neuhauser H, Leopold M, von Brevern M, Arnold G, Lempert T. The interrelations of migraine, vertigo, and migrainous vertigo. Neurology. 2001 Feb 27;56(4):436-41. doi: 10.1212/wnl.56.4.436. PMID 11222783
- [Background] Formeister EJ, Rizk HG, Kohn MA, Sharon JD. The Epidemiology of Vestibular Migraine: A Population-based Survey Study. Otol Neurotol. 2018 Sep;39(8):1037-1044. doi: 10.1097/MAO.0000000000001900. PMID 30020261